CLINICAL TRIAL: NCT00398736
Title: A Non-invasive Approach to the Assessment of Volume Status in Mechanically Ventilated Septic Patients.
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Other Study IDs: Caval vein sonography
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Presence of severe sepsis and septic shock, mechanical ventilation
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: sonographic measurement of inferior caval vein diameter

SUMMARY:
To evaluate the use of sonographic inferior caval vein assessment in mechanically ventilated septic patients.

Volume assessment in mechanically ventilated patients with inflammation is of major importance to guide fluid therapy. The researchers investigated whether measurement of caval vein diameter correlates with invasively assessed volume-based hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90
* presence of severe sepsis and septic shock
* invasive hemodynamic monitoring using the picco system

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Dr. Schefold, MD, Principal Investigator — Charite University Medicine